CLINICAL TRIAL: NCT06233565
Title: Dexamethasone vs. Dexmedetomidine for Popliteal Nerve Block in Pain Management After Pediatric Ankle and Foot Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/2024
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-04

CONDITIONS: Foot Injuries and Disorders; Ankle Injuries and Disorders
MeSH Terms: conditions — Foot Injuries; Disease; Ankle Injuries | interventions — Sodium Chloride; Dexamethasone; Calcium Dobesilate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.9%sodium chloride
- Dexamethasone (Active Comparator): 0.2% ropivacaine + 0.1mg/kg Dexamethasone for popliteal nerve block
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Active Comparator): 0.2% ropivacaine + 0.1ug/kg Dexmedetomidine for popliteal nerve block
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: 0.9%sodium chloride — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the popliteal nerve block
  Other Names: placebo
  Arms: Placebo
Drug: Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the popliteal nerve block
  Other Names: desamethasone
  Arms: Dexamethasone
Drug: Dexmedetomidine — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1ug/kg Dexmedetomidine for the popliteal nerve block
  Arms: Dexmedetomidine

SUMMARY:
Effect of perineurial dexamethasone and dexmedetomidine on popliteal nerve block duration for pediatric, ankle or foot surgery

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineurial Dexamethasone and Dexmedetomidine on erector spinal plane block duration for pediatric, idiopathic scoliosis surgery.

After scoliosis surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone or Dexmedetomidine, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone and Dexmedetomidine use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare perineural Dexamethasone and Dexmedetomidine. Group 2 has dexamethasone doses of 0.1mg/kg, and group 3 has 0,1ug/kg Dexmedetomidine added to the local anesthetic.

The investigator aims to find a dexamethasone or dexmedetomidine that covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* all children scheduled for ankle or foot surgery
* aged > 3 months < 7 years

Exclusion Criteria:

* age < 3 months
* age > 7 years
* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use
* chronic pain

Ages: 3 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | [Time Frame: 4 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | [Time Frame: 6 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | [Time Frame: 8 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | [Time Frame: 12 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | [Time Frame: 24 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | [Time Frame: 48 hours after surgery]
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
NLR | 24 and 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 24 and 48 hours after surgery
  Platelet-to-lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (2):
- Poland (2):
  - Poznan University of Medical Sciences, Poznan, Poznań
  - Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reysner T, Pietraszek P, Shadi M, Musielak B, Kowalski G, Daroszewski P, Reysner M. Effect of perineural dexamethasone versus dexmedetomidine as adjuvants to ropivacaine on analgesic duration in pediatric popliteal sciatic nerve blocks: a randomized, triple-blinded, placebo-controlled trial. Reg Anesth Pain Med. 2025 Oct 2:rapm-2025-107096. doi: 10.1136/rapm-2025-107096. Online ahead of print. PMID 41043950